CLINICAL TRIAL: NCT04780776
Title: Evaluating the Effect of SOLIUS UV Light Source in Improving Serum Levels of 25-hydroxyvitamin D in Vitamin D Deficient/ Insufficient Adults of Various Skin Types
Brief Title: Evaluating the Effect of SOLIUS UV Light Source in Improving Vitamin D Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-40850
Record Dates: First submitted 2021-02-26; First posted 2021-03-04 (Actual); Results first posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Vitamin D Deficiency; Vitamin D Insufficiency
Keywords: Vitamin D; Ultraviolet B radiation; SOLIUS System
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- UVB treatment arm (Experimental): The treatment group will first undergo an evaluation of each individual's sensitivity to the SOLIUS System UVB using the device titration system for the first 5 weeks. Once the UVB dose is determined during the 5 weeks, the subjects will be enrolled in a 16-week study where they will be exposed to their individualized dose.
  Interventions: Device: UVB treatment
- Sham comparator arm (Sham Comparator): The sham comparator group will undergo the procedures as the treatment group with the exception that the SOLIUS System will only be turned on to emit visible radiation.
  Interventions: Device: Sham comparator

INTERVENTIONS:
Device: UVB treatment — 5 weeks of UVB titration to determine individual's UVB sensitivity followed by 16 weeks of UVB exposure intervention
  Arms: UVB treatment arm
Device: Sham comparator — 5+16 weeks of visible light exposure
  Arms: Sham comparator arm

SUMMARY:
The aim of this study is to evaluate the safety and effectiveness of the SOLIUS System in improving serum levels of 25-hydroxyvitamin D in vitamin D deficient/ insufficient adults of various skin types.

The investigators will conduct a double-blinded randomized clinical trial in 100 adults to compare the changes in serum 25-hydroxyvitamin D levels between subjects who received and do not receive weekly exposures to Ultraviolet B Radiation (UVB) generated by the SOLIUS System for 16 weeks.

DETAILED DESCRIPTION:
Study enrollment

Approximately 100 healthy adults will be enrolled ages 22 or older; both sexes, for vitamin D deficiency screening in order to enroll 80 adults with vitamin D deficiency/insufficiency (serum 25-hydroxyvitamin D <30 ng/mL). Participants will be randomized 1:1 into two groups: 40 adults for treatment arm who will receive weekly exposures of ultraviolet radiation generated by the SOLIUS System, and 40 adults for sham comparator arm.

Study procedure

The treatment group that will be exposed to the SOLIUS System will first undergo an evaluation of each individual's sensitivity to the SOLIUS System UVB using the device titration system for the first 5 weeks. Once the UVB dose is determined during the 5 weeks, the subjects will be enrolled in a 16-week study where they will be exposed to their individualized dose. For the sham comparator group, they will undergo the procedures as the treated group with the exception that the SOLIUS System will only be turned on to emit visible radiation. At these visits, each subject assigned into both groups will be asked questions about consumption of vitamin D, sun exposure, and whether he/she has had any adverse changes in his/her health. Serum 25-hydroxyvitamin D levels will be measured at baseline and monthly, and the levels will be analyzed to compare between those who receive and who do not receive the UVB radiation intervention for baseline and during the 16-week treatment period. After the 16-week intervention, participants will be asked to return to the study site weekly for measurement of serum 25-hydroxyvitamin D for 4 weeks. Serum 25(OH)D levels will be determined using the Liquid Chromatography with tandem mass spectrometry (LC/MS/MS) method. Safety will be monitored by interviewing the participants after each UVB exposure for any adverse events, including erythema or any other skin reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 22 years old
2. Male or Female
3. Skin Type I-VI
4. Women of child bearing potential must be on birth control and not pregnant based on a negative pregnancy test at baseline.
5. Ability and Willingness to give informed consent and comply to protocol requirements
6. Serum total 25(OH)D < 30 ng/mL at the screening

Exclusion Criteria:

1. Ongoing treatment with supplemental or pharmacological doses of vitamin D, vitamin D metabolites or analogues
2. Pregnant
3. History of underlying photosensitivity
4. Use of medications that cause a photosensitivity reaction (including but not limited to): tetracycline, tretinoin, amiodarone, doxycycline, naproxen, diphenhydramine, methotrexate, and hydrochlorothiazide
5. History of skin cancer
6. Plan to received significant sun exposure below the 33rd parallel during study
7. Used tanning or phototherapy devices within the last 30 days
8. Vitamin D supplement use of more than 600 IUs daily
9. Systemic steroids use
10. H1 antihistamine use in the last 7 days
11. Diagnosed with light allergies (including but not limited to): actinic prurigo, polymorphous light eruption, or solar urticaria
12. Diagnosed with light sensitivities (including but not limited to): protoporphyria, photodermatitis, xeroderma pigmentosum, lupus erythematosus, chronic actinic dermatitis, or UV-sensitive syndrome

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Holick, MD PhD, Principal Investigator — Boston University
Locations (1):
- BU School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screened adults with vitamin D deficiency or insufficiency were selected for the study and randomized into the two study arms.
Groups:
- UVB Treatment Arm: Participants receive ultraviolet B radiation (UVB) exposure from the SOLIUS System.
- Sham Comparator Arm: Participants receive blue/violet light exposure from the SOLIUS System.
Period: Titration Week 1-5
Arm/Group | UVB Treatment Arm | Sham Comparator Arm
Started | 35 | 34
Completed | 33 | 26
Not Completed | 2 | 8
Not completed — Lost to Follow-up | 2 | 8
Period: Treatment Week 6-21
Arm/Group | UVB Treatment Arm | Sham Comparator Arm
Started | 33 | 26
Completed | 29 | 22
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4
Period: Follow up Week 22-25
Arm/Group | UVB Treatment Arm | Sham Comparator Arm
Started | 29 | 22
Completed | 27 | 20
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UVB Treatment Arm | Sham Comparator Arm | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.09 (10.78) | 34.44 (11.40) | 34.26 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 12 | 13 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8 | 3 | 11
  Black | 6 | 13 | 19
  Black- Cape Verde | 1 | 0 | 1
  Black- Hispanic | 1 | 0 | 1
  Black- Multirace | 0 | 1 | 1
  Hispanic | 4 | 4 | 8
  Hispanic- White | 1 | 0 | 1
  Hispanic- Multirace | 1 | 0 | 1
  Multirace | 0 | 1 | 1
  White | 13 | 12 | 25
Region of Enrollment [Number; unit: participants]
  United States | 35 | 34 | 69
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick Skin Types: Type II [Fair skin, blue eyes, Burns easily, tans poorly]; Type III [Darker white skin, Tans after initial burn]; Type IV [Light brown skin, Burns minimally, tans easily]; Type V [Brown skin, Rarely burns, tans darkly easily].
  Participants
    Skin Type II/III | 30 | 30 | 60
    Skin Type IV/V | 5 | 4 | 9
Screening 25(OH)D Levels [Mean (Standard Deviation); unit: ng/mL] | 20.57 (5.30) | 19.71 (5.16) | 20.41 (5.21)

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum 25-Hydroxyvitamin D [25(OH)D]
Description: This outcome measures the change in serum 25-hydroxyvitamin D [25(OH)D] concentrations in participants from Week 1 to the end of the intervention period Week 21.
Time Frame: Week 1, Week 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | UVB Treatment Arm | Sham Comparator Arm
Number analyzed (Participants) | 27 | 20
ng/mL | 10.14 (7.5) | -2.3 (4.9)

2. Primary Outcome: Distribution of Participants by Vitamin D Deficiency Categories at Week 1
Description: The three vitamin D categories are defined as: Deficient - <20 ng/mL 25(OH)D, Insufficient - 21-29 ng/mL 25(OH)D, Sufficient - 30-100 ng/mL 25(OH)D.
Time Frame: Week 1
Population: Only participants who completed the treatment are analyzed (27 in the treatment and 20 in the control arm).
Measure: Count of Participants; unit: Participants
Arm/Group | UVB Treatment Arm | Sham Comparator Arm
Number analyzed (Participants) | 27 | 20
Participants
  Deficient | 19 | 9
  Insufficient | 6 | 10
  Sufficient | 2 | 1

3. Primary Outcome: Distribution of Participants by Vitamin D Deficiency Categories at Week 21
Description: as for outcome 2
Time Frame: Week 21
Population: Only participants who completed the treatment are analyzed (27 in the treatment and 20 in the control arm).
Measure: Count of Participants; unit: Participants
Arm/Group | UVB Treatment Arm | Sham Comparator Arm
Number analyzed (Participants) | 27 | 20
Participants
  Deficient | 3 | 16
  Insufficient | 13 | 4
  Sufficient | 11 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- UVB Treatment Arm: Participants receive ultra violet radiation (UVB) exposure from the SOLIUS System.
Arm/Group | UVB Treatment Arm | Sham Comparator Arm
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 23/35 | 13/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UVB Treatment Arm (N=35) | Sham Comparator Arm (N=34)
Redness (Skin and subcutaneous tissue disorders) | 12 | 6
Itchiness (Skin and subcutaneous tissue disorders) | 8 | 4
Tenderness (Skin and subcutaneous tissue disorders) | 4 | 4
Darkening/tanning (Skin and subcutaneous tissue disorders) | 4 | 2
Tightness (Skin and subcutaneous tissue disorders) | 4 | 2
Dryness (Skin and subcutaneous tissue disorders) | 3 | 0
Peeling (Skin and subcutaneous tissue disorders) | 2 | 0
Discomforts (Skin and subcutaneous tissue disorders) | 1 | 2
Sensitivity (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT04780776/Prot_SAP_000.pdf